CLINICAL TRIAL: NCT05338931
Title: An Open-label, Single-arm, Multi-center, Phase I/II Study to Evaluate the Safety, Tolerability, and Efficacy of AT101 (Anti-CD19 Chimeric Antigen Receptor T Cell) in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Safety, Tolerability, and Efficacy of AT101 in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbClon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AbClon
Record Dates: First submitted 2022-04-01; First posted 2022-04-21 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: B-cell Non Hodgkin Lymphoma
Keywords: Anti-CD19 Chimeric Antigen Receptor T cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — gossypol acetic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AT101(Anti-CD19 Chimeric Antigen Receptor T cell) (Experimental): Anti-CD19 Chimeric Antigen Receptor T cell
  Interventions: Drug: AT101(Anti-CD19 Chimeric Antigen Receptor T cell)

INTERVENTIONS:
Drug: AT101(Anti-CD19 Chimeric Antigen Receptor T cell) — Anti-CD19 Chimeric Antigen Receptor T cell
  Other Names: AT101

SUMMARY:
Determine MTD based on the safety and tolerability of AT101 and the RP2D for patients with recurrent or non-reactive B-cell NHL.

DETAILED DESCRIPTION:
Determine the maximum tolerant dose (MTD) based on the safety and tolerability of AT101 and the recommended dose 2 dose (RP2D) in phase 2 trials for patients with recurrent or non-reactive B cell non-Hodgkin lymphoma (B-cell NHL).

ELIGIBILITY:
Inclusion Criteria:

* B cell non-Hodgkin lymphoma based on WHO classification 2017
* incompatible with existing standard therapies or have had disease progression, and whose standard therapies do not currently have available standard therapies due to reasons such as intolerance/inadequacies or rejection
* The Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* adequate hematological, kidney, liver, lung, heart and bone marrow function without blood transfusion within two weeks prior to screening
* Those with a minimum life expectancy of 12 weeks or more
* In women with childbearing, clinical response tests (serum- or ure-hCG) were negatively identified during this trial
* Those who have agreed in writing to participate voluntarily in this trial

Exclusion Criteria:

* Those who have previously had a history of treating homologic autologous hemoblastitis (allogeneic HSCT)
* At101/adcidmilisers, anticancer chemotherapy/adcidms for lymphodeletion or those who are hypersensitive to tocilizumab
* Those who cannot take autologous blood
* Those who have received chemotherapy or radiotherapy, excluding lymphodeletion, within two weeks prior to IP administration
* Persons who have not been recovered (CTCAE grade ≤1 or baseline) due to previous treatment
* Those who have identified a condition that, at the test's discretion, may affect safety and validation during the trial period.
* Those who have identified the following forces at the time of screening:

  1. Those who have been clinically aware of heart disease within 6 months prior to screening
  2. Those identified as thromboembolic disease, pulmonary embolism or bleeding bleeding diatheses within 6 months prior to screening
  3. Those who have identified a history of malignant tumors other than B-cell non-Hodgkin's lymphoma within five years prior to screening
  4. Those who have undergone major surgery within 4 weeks prior to screening
  5. Those who have undergone non-critical surgery within two weeks prior to screening
* Childbearing women or men who do not have the will to use effective contraception for a longer period of time, either 12 months after clinical trial period and AT101 administration or when AT101 in the body is not identified
* Those who have been administered or applied to other IP/ID within 4 weeks of screening
* Those who are addicted to alcohol and/or medication
* Those who are unfit or unable to participate in this trial when judged by PI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2030-03-15 (Estimated); Study Completion 2030-09-15 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerant dose (MTD) and Recommended Phase 2 Dose (RP2D) | 28 days
  Phase I: Tolerability of AT101 and the recommended dose 2 dose (RP2D) in phase 2 trials
Overall response rate (ORR) by Independent assessment | 5 years
  Phase II: Proportion of subjects whose best overall response in tumor evaluation was evaluated as a complete response or a partial response

SECONDARY OUTCOMES:
Overall response rate (ORR) by Investigator assessment | 5 years
  Proportion of subjects whose best overall response in tumor evaluation
Duration of overall response (DOR) | 5 years
  Time from first response (CR or PR) to the date of initial objectively documented progression
Overall survival(OS) | 5 years
  Time from randomization to death
Progression free survival (PFS) | 5 years
  Time from randomization to disease progression or death
Time to response (TTR) | 5 years
  Time from randomization to CR or PR
Event free survival (EFS) | 5 years
  Time from randomization to progression, subsequent chemotherapy or death
Incidence of adverse Event | 5 years
Peak concentration (Cmax) of AT101 | 5 years
Area under the concentration versus time curve (AUC) of AT101 | 5 years
AT101 transgene expression | 5 years
Replication-competent lentivirus (RCL) as Assessed by quantitative polymerase | 5 years

OTHER OUTCOMES:
Concentration of cytokines | 5 years
CD19 expression | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Deok-hyun Yoon, Principal Investigator — Asan Medical Center, 88, Olympic-ro 43-gil, Songpa-gu, Seoul, South Korea
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Zhang Y, Patel RP, Kim KH, Cho H, Jo JC, Jeong SH, Oh SY, Choi YS, Kim SH, Lee JH, Angelos M, Guruprasad P, Cohen I, Ugwuanyi O, Lee YG, Pajarillo R, Cho JH, Carturan A, Paruzzo L, Ghilardi G, Wang M, Kim S, Kim SM, Lee HJ, Park JH, Cui L, Lee TB, Hwang IS, Lee YH, Lee YJ, Porazzi P, Liu D, Lee Y, Kim JH, Lee JS, Yoon DH, Chung J, Ruella M. Safety and efficacy of a novel anti-CD19 chimeric antigen receptor T cell product targeting a membrane-proximal domain of CD19 with fast on- and off-rates against non-Hodgkin lymphoma: a first-in-human study. Mol Cancer. 2023 Dec 9;22(1):200. doi: 10.1186/s12943-023-01886-9. PMID 38066564